CLINICAL TRIAL: NCT07192120
Title: A Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of MHB048C for Injection in Patients With Advanced Solid Tumors
Brief Title: A Study of MHB048C in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MHB048C-A-101
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: mCRPC (Metastatic Castration-resistant Prostate Cancer); Advanced Malignant Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MHB048C (Phase I: Dose escalation) (Experimental): There are seven escalating dose cohorts.
  Interventions: Drug: MHB048C for Injection
- MHB048C (Phase II: Dose expansion) (Experimental): The recommended dose from the dose-escalation stage and other potential doses will be further explored.
  Interventions: Drug: MHB048C for Injection

INTERVENTIONS:
Drug: MHB048C for Injection — IV administration of MHB048C Q2W or Q3W; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.

SUMMARY:
This is a first-in-human, open-label, multicenter Phase I/II study of MHB048C in patients with advanced solid tumors. The study was designed to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of MHB048C monotherapy.

DETAILED DESCRIPTION:
This first-in-human clinical trial of MHB048C comprises two parts: a dose escalation phase and a dose expansion phase. The dose escalation phase is an open-label, multicenter study including dose escalation and PK expansion cohorts. The primary objectives are to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of MHB048C in patients with advanced solid tumors, and to determine the maximum tolerated dose (MTD). In this phase, additional patients may be enrolled in the PK expansion part at dose levels that have completed DLT (dose-limiting toxicity) evaluation.

Based on the safety, PK, and preliminary efficacy data from the completed DLT-evaluated dose levels, the sponsor will initiate the dose expansion phase. This phase is an open-label, multicenter, multi-cohort study designed to further evaluate the safety and efficacy of MHB048C monotherapy in patients with mCRPC or other types of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agrees to participate in the study and signs the informed consent form.
2. Age ≥ 18 years, no restriction on gender.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Estimated life expectancy ≥ 3 months.
5. Histologically or cytologically confirmed advanced solid tumors that are refractory to standard therapy, intolerant to standard therapy, or have no standard treatment options.
6. At least one measurable lesion per RECIST v1.1 criteria or one bone.
7. Adequate bone marrow reserve and organ function. -

Exclusion Criteria:

1. History of ≥2 primary malignancies within 5 years prior to informed consent.
2. Received chemotherapy within 3 weeks, radiotherapy within 4 weeks, or biologic, endocrine, or immunotherapy within 4 weeks before first study dose.
3. Medication of other unmarketed investigational drugs or therapies within 4 weeks before the first dose of investigational drug.
4. Brain metastases, bone marrow metastases, leptomeningeal disease, brainstem metastases, or spinal cord compression.
5. Severe bone damage caused by bone metastasis of prostate cancer.
6. Has adverse reactions from previous anti-tumor treatment that have not recovered to ≤ CTCAE 5.0 Grade 1.
7. Severe lung disease affecting pulmonary function.
8. Vaccinated within 4 weeks before dosing.
9. Active systemic infection requiring treatment within 7 days before dosing.
10. Serious cardiovascular or cerebrovascular diseases.
11. Uncontrolled third-space effusions not suitable for enrollment.
12. Significant bleeding, bleeding tendency, or non-healing wounds within 1 month before first dose.
13. Known hypersensitivity or delayed allergic reaction to the investigational product or its components.
14. Drug abuse or other medical/psychiatric condition that may interfere with study participation or results.
15. Known alcohol or drug dependence.
16. Pregnant or breastfeeding women, or individuals planning to conceive. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
(Dose-Escalation Stage): Dose-Limiting Toxicity (DLT) and Maximum tolerated dose (MTD) for MHB048C | Up to day 21 from the first dose for Q3W administration.
  To determine the MTD for further evaluation of IV administration of MHB048C monotherapy in subjects with advanced solid tumors.
(Dose-Expansion Stage): Objective tumor response (ORR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  To determine the recommended Phase II dose (RP2D) of MHB048C for the treatment of selected patients with advanced solid tumors based on the safety and efficacy results from all enrolled subjects.

SECONDARY OUTCOMES:
ORR determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of CR and PR (Confirmed CR/PR assessment require at least 1 repeat).
Duration of response (DOR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  DoR was defined as the period from the first occurrence of CR or PR to PD or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].
Disease control rate (DCR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks); SD shall be assessed at least 5 weeks after the first dose].
Radiographic Progression-free survival (rPFS) determined by investigators according to PCWG3 | Baseline up until radiographic progression on bone lesion, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  rPFS was defined as the time from random assignment (dose expansion stage) or first dose (dose escalation stage) to radiographic progression on bone lesion.
Overall survival (OS) | Baseline up until death up to approximately 5 years
  OS was defined as the time from random assignment or first dose to death from any cause.
Incidence and severity of adverse events (AEs), serious adverse events (SAEs), AEs leading to treatment suspension, discontinuation | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years.
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0].
Pharmacokinetic (PK) parameters of total antibody, ADC, and free toxin at various time points | From pre-dose to 22 days after the first dose.
  The PK parameters at different time points include: Area Under the Concentration-Time Curve (AUC)
Pharmacokinetic (PK) parameters of total antibody, ADC, and free toxin at various time points | From pre-dose to 22 days after the first dose.
  The PK parameters at different time points include: Maximum Plasma Concentration (Cmax)
Immunogenicity | From pre-dose to 30 days post end of treatment.
  Proportion of subjects who develop anti-MHB048C antibodies (ADA).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No